CLINICAL TRIAL: NCT00064831
Title: The Effect of Black Cohosh Extract on the Human Breast
Brief Title: Black Cohosh Extract in Postmenopausal Breast Health
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Edward Sauter, MD, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21AT001102-01 (NIH); SauterE
Record Dates: First submitted 2003-07-14; First posted 2003-07-15 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Menopause; Hot Flashes
Keywords: estrogen stimulation; relief of hot flashes; nipple aspirate fluid; body fluid levels of black cohosh
MeSH Terms: conditions — Hot Flashes | interventions — black cohosh root extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Black Cohosh Extract (BCE)

SUMMARY:
The purpose of the study is to determine if black cohosh extract (BCE) administration in symptomatic postmenopausal women results in estrogenic stimulation of the breast, as determined by estradiol, pS2, FSH, LH, and PSA levels in nipple aspirate fluid.

DETAILED DESCRIPTION:
As in Brief Summary

ELIGIBILITY:
* Postmenopausal females
* 20 months since any breastfeeding
* Active postmenopausal symptoms, i.e., hot flashes
* At least 6 months since last menstrual period or have had a hysterectomy with both ovaries removed
* Able to make 4 visits during the trial to the study clinic in Columbia, Missouri

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73
Dates: Start 2003-07; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Sauter, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States